CLINICAL TRIAL: NCT05410340
Title: Brain Activation and Oxygenation Through Reflex Locomotion Therapy (Vojta) and Massage in Preterm Infants
Brief Title: EEG and NIRS in Preterm Infants
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Rocío Llamas-Ramos, Associate Professor, University of Salamanca
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: EEGNIRS2022
Record Dates: First submitted 2022-05-28; First posted 2022-06-08 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Premature Birth
Keywords: Preterm; Premature; Infant; Baby; Child
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Invesigator will not know which infants are premature or not
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Preterm group 1 (Active Comparator): To analize the brain activation and oxigenation using the Vojta Therapy
  Interventions: Other: Vojta Therapy
- Preterm Group 2 (Active Comparator): To analize the brain activation and oxigenation using massotherapy
  Interventions: Other: Massotherapy
- Term group 1 (Placebo Comparator): To analize the brain activation and oxigenation using the Vojta Therapy
  Interventions: Other: Vojta Therapy
- Term group 2 (Placebo Comparator): To analize the brain activation and oxigenation using massotherapy
  Interventions: Other: Massotherapy

INTERVENTIONS:
Other: Vojta Therapy — Minimal digital pressure at costal level to assess the activation and oxygenation occurring at the cerebral level
  Arms: Preterm group 1; Term group 1
Other: Massotherapy — Baby body massage with gliding
  Arms: Preterm Group 2; Term group 2

SUMMARY:
Experimental cross-sectional study of a single application (vojta therapy or massage) in preterm and non-preterm infants to test whether there are differences in brain activation and oxygenation that occur with both techniques between term and preterm infants.

Secondly, the brain activation and oxygenation produced by both physiotherapy techniques will be tested separately to establish comparisons between the two groups.

Finally, between 3 - 6 months, we will analyse whether there are changes in gaze fixation (eye tracker) in the 4 study arms to see if there are differences between term and preterm infants but also the differences between the immediate effectiveness of both techniques.

ELIGIBILITY:
Inclusion Criteria:

* term and preterm babys
* first month after birth

Exclusion Criteria:

* intrumental delivery
* pathology associated

Ages: 7 Days to 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2024-08-03 (Actual); Primary Completion 2024-10-02 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
EEG (Alpha, Beta, Theta) | Change from Baseline brain activation at 3 months
  Brain activation
NIRS | Change from Baseline brain oxigenation at 3 months
  Brain oxigenation

SECONDARY OUTCOMES:
Eye tracker | Change from Baseline gaze fization at 6 months
  Gaze fixation

CONTACTS AND LOCATIONS:
Locations (1):
- University of Salamanca, Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: Undecided